CLINICAL TRIAL: NCT01933256
Title: A Randomized, Double-blind, Placebo-controlled Study of the Effect of 49 Days of Treatment With Repeated Subcutaneous Doses of HIP2B to Assess Safety, Tolerability and Measures of Islet β-cell Function in Subjects With Type 2 Diabetes Mellitus Treated With Metformin
Brief Title: Study of Subcutaneous Doses of HIP2B in Subjects With Type 2 Diabetes Mellitus Treated With Metformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CureDM (Industry)
Collaborators: Profil Institute for Clinical Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: TDU1156-002
Record Dates: First submitted 2013-08-05; First posted 2013-09-02 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; HIP2B; Placebo; islet β cell
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 600mg HIP2B (Experimental): 600mg HIP2B
  Interventions: Drug: HIP2B
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 400mg HIP2B (Experimental): 400mg HIP2B
  Interventions: Drug: HIP2B

INTERVENTIONS:
Drug: HIP2B
  Arms: 400mg HIP2B; 600mg HIP2B
Drug: Placebo
  Arms: Placebo

SUMMARY:
HIP2B is being developed for the treatment of type 1 and type 2 diabetes mellitus.

The purpose of this study is to investigate the safety and tolerability of repeat doses of HIP2B in subjects with type 2 diabetes mellitus. The study will also assess whether islet β-cell number and function will increase over time in response to repeat HIP2B injections.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 30 to 65 years, inclusive
* Males and females
* Diagnosis of type 2 diabetes mellitus prior to screening meeting the following criteria:

  1. Body mass index <45 kg/m2
  2. HbA1c value of > 6.5 to <9.5%
  3. C-peptide ≥1.0 ng/mL
  4. On a stable dose of metformin for 12 weeks
* Ability to provide written informed consent and be willing to comply with scheduled visits, treatment plan, laboratory tests and other study procedures

Exclusion Criteria:

* History of any of the following: type 1 diabetes mellitus, diabetic ketoacidosis, an episode of severe hypoglycemia (defined as a change in mental status requiring assistance) during the prior 30 days
* FPG >260 mg/dL at time of randomization
* Current or chronic use (within past 12 weeks) of insulin, or insulin secretagogues including: sulfonylureas, GLP-1 analogs, DPP-4 inhibitors, meglitinides, α-glucosidase inhibitors, pioglitazone, or rosiglitazone
* Glomerular filtration rate (GFR) <60 as calculated using the Modified Diet in Renal Disease equation at screening
* ALT, AST or total bilirubin > 2 X ULN
* Serum amylase concentration > 1.5XULN or serum lipase concentration >2XULN
* Positive test result for glutamic acid decarboxylase antibodies (GADA).
* The presence of a clinically significant abnormality on resting electrocardiogram (ECG)
* Positive HIV, hepatitis B (HBsAg), or positive hepatitis C (HCV Ab) test at screening
* History of clinically significant renal, hepatic, cardiovascular, neurological, or gastrointestinal disease that could impact patient safety in the investigator's opinion
* Serum triglycerides >500 mg/dL
* Presence or history of cancer within the past 5 years with the exception of adequately treated localized basal cell skin cancer or in situ uterine cervical cancer
* History of weight loss > 5% in the 8 weeks prior to randomization or subject is on a weight loss program and is not in the maintenance phase
* Use of any weight loss medication within 8 weeks of randomization
* Uncontrolled hypertension defined as blood pressure >160/100 mmHg, using an appropriately sized cuff, at rest
* History or evidence of multiple organ autoimmune disorders
* History of thyroid dysfunction other that hypothyroidism treated with stable dose of thyroid hormone and euthyroid at screening
* History or presence of acute or chronic pancreatitis or symptomatic recurrent gallstones
* Has undergone surgery within 6 months of screening or plans to undergo surgery during the study period
* Use of parenterally administered proteins or antibodies within 12 weeks of screening. (Note: Influenza vaccine will be allowed.)
* Prior exposure to any investigational agent or participation in an investigational trial within 30 days prior to Day 1
* Blood loss or blood donation >500 ml in the 2 months prior to screening.
* Use of systemic long-acting corticosteroids within two months or prolonged use (more than one week) of other systemic corticosteroids or inhaled corticosteroids (if daily dosage is >1000 mcg equivalent beclomethasone) within 30 days prior to screening visit.
* Drugs with the potential to affect (either increasing or decreasing) endogenous insulin secretion or insulin sensitivity including corticosteroids (as detailed above), β-adrenergic blockers, beta-adrenergic agonists, quinine, thiazide or thiazide-like diuretics, calcineurin inhibitors, niacin, anti-psychotic or antidepressant drugs, somatostatin analogs, growth hormone, weight-reducing drugs (e.g. orlistat, phentermine and topiramate extended-release, lorcaserin). Stable doses of agents commonly required by subjects with T2DM including angiotensin converting enzyme inhibitors, angiotensin II receptor blockers, statins, fibrates, and aspirin (<100 mg daily) will be permitted at the discretion of the investigator.
* A serious adverse reaction or hypersensitivity to any drug, unless reaction deemed irrelevant to the study by the investigator and sponsor.
* History of alcohol abuse or drug abuse within the previous 12 months. No history of medical or recreational use of marijuana within previous 12 months.
* A history of smoking more than one-half a pack of cigarettes per day within last 12 months
* History of stroke, transient ischemic attack or myocardial infarction within 6 months prior to screening.
* History of New York Heart Association Class II-IV heart failure prior to screening.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of repeat doses of HIP2B in subjects with type 2 diabetes mellitus. | Adverse Events / vitals are monitored at each study visit between Days -9 and 84.
  Safety evaluations will include clinical observation and adverse event (AE) reporting; evaluation of the injection site, physical examination, vital signs; electrocardiograms (ECGs), hematology, chemistry panels (inclusive of expanded markers of liver function), dipstick urinalysis (microscopic evaluation if dipstick positive), amylase, LDH.

SECONDARY OUTCOMES:
Glucose-stimulated insulin secretion. | IVGTT performed on Day -8 and Day 49. GGI performed on Day -1, Day 25 and Day 46.
  First-phase insulin response will be assessed (a) as the incremental insulin peak (above baseline) after glucose injection during the IVGTT and (b) as the incremental insulin area obtained over 10 min; incremental area under the curve (AUC) during the GGI will be calculated for insulin and C-peptide.

OTHER OUTCOMES:
Pre-hepatic insulin secretion rate. | GGI used for assessments is performed on Day -1, Day 25 and Day 46.
  The pre-hepatic insulin secretion rate will be calculated based on deconvolution of peripheral C-peptide concentrations during GGI using the method described by Hovorka et al.
Change in β-cell responsiveness. | GGI measured on Day-1, Day 25 and Day 46.
  Change in β-cell responsiveness will be assessed by comparing the slopes of the change of plasma insulin against glucose before and after treatment.
PK parameters of HIP2B after single and repetitive dosing. | PK testing done on Day 1 and Day 46 at pre-dose, 15 and 30min, 1 and 2 hours post dose.
  PK parameters of HIP2B: e.g. Cmax, Tmax, AUC (0.t), AUC(0-∞), CL/F, V/F, t½.
Pharmacodynamic (PD) effects of repeat doses of HIP2B on measures of glycemic control and β-cell function | Assessments completed at screening, Days -9, -8, -2, -1, 1, 7, 14, 21, 24, 28, 42, 45, 46, 48, 49, 61, 68, and 84.
  Pharmacodynamic (PD) effects of repeat doses of HIP2B on measures of glycemic control and β-cell function including fasting plasma glucose, fasting C-peptide, fasting proinsulin/insulin ratio and HOMA-B; glycated albumin, HbA1c, and 7-point glucose profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Hompesch, MD, Principal Investigator — Profil Institute for Clinical Research, Inc.
Locations (1):
- Profil Institute for Clinical Research, Inc., Chula Vista, California, United States